CLINICAL TRIAL: NCT03018639
Title: Impact of Therapist Change After Initial Contact and Traumatic Burden on Dropout in a Naturalistic Sample of Inpatients With Borderline Pathology Receiving Dialectical Behavior Therapy
Brief Title: Impact of Therapist Change on Dropout in a Naturalistic Sample of Inpatients With Borderline Pathology Receiving DBT
Status: Completed | Type: Observational
Sponsor: Evangelisches Krankenhaus Bielefeld gGmbH (Other)
Responsible Party: Principal Investigator, Carolin Steuwe, Research Associate, Evangelisches Krankenhaus Bielefeld gGmbH
Other Study IDs: DBT_dropout
Record Dates: First submitted 2017-01-09; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Borderline Personality Disorder; PostTraumatic Stress Disorder; Psychotherapy; Dropout
MeSH Terms: conditions — Borderline Personality Disorder; Stress Disorders, Post-Traumatic | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dialectical Behavior Therapy: The program's purpose is to help patients achieve the following therapeutic goals: (1) reduction of suicidal behaviors, (2) reduction of therapy-interfering behaviors, and (3) other risky or destabilizing behaviors. Standard DBT aims to achieve these goals by (1) conveying behavioral capabilities (skills), (2) motivation for applying these skills, (3) generalization of learned skills to the patient's natural environment, (4) structuring the treatment environment to reinforce functional behavior, and (5) conveying therapeutic resources and motivation to effectively treat patients with BPD.
  Interventions: Behavioral: Dialectical Behavior Therapy

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy — DBT is a cognitive-behavioral treatment program that was developed to treat suicidal Patients with BPD (Linehan, 1993).

SUMMARY:
Participants with Borderline pathology (≥ 3 DSM-IV-criteria) receiving an inpatient Dialectical Behavior Therapy (DBT) program completed a quality assurance questionnaire set assessing demographic information and pretreatment psychopathology during the days of their inpatient stay. Beyond that, changes of therapists were documented.

ELIGIBILITY:
Inclusion Criteria:

* three or more criteria for BPD as defined by DSM-IV (Borderline Personality characteristics; BPC)

Exclusion Criteria:

* inability to contract and consent,
* other severe mental disorders (bipolar disorder, acute psychosis),
* current alcohol,
* illicit or not prescribed drug use,
* simultaneous participation in other treatment studies,
* pregnancy or breastfeeding,
* an inability to negotiate a non-suicide agreement,
* ongoing traumatic contact with the perpetrator, and
* a Body Mass Index < 16.5.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study, all patients aged from 18 to 65, discharged from our personality disorder inpatient unit between December 2012 and August 2016, and fulfilling three or more criteria for BPD as defined by DSM-IV (Borderline Personality characteristics; BPC) were considered (n = 89).
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2012-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Dropout | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Driessen, Study Director — Research Department, Ev. Krankenhaus Bielefeld
Locations (1):
- Research Department, Bielefeld, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steuwe C, Berg M, Driessen M, Beblo T. Impact of therapist change after initial contact and traumatic burden on dropout in a naturalistic sample of inpatients with borderline pathology receiving dialectical behavior therapy. Borderline Personal Disord Emot Dysregul. 2017 Jun 22;4:14. doi: 10.1186/s40479-017-0067-3. eCollection 2017. PMID 28649383